CLINICAL TRIAL: NCT05766098
Title: Caratterizzazione Del Profilo Mutazionale Nel Tumore Papillare Della Tiroide Tramite Tecnologia Mass-ARRAY
Brief Title: Definition of Mutational Profile of Papillary Thyroid Tumors by Mass-ARRAY
Acronym: PTC-ARRAY
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 05C825
Record Dates: First submitted 2023-02-28; First posted 2023-03-13 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — papillary thyroid tumor tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with papillary thyroid cancer
  Interventions: Genetic: Genotyping

INTERVENTIONS:
Genetic: Genotyping — Characterization of genetic profile of tumor tissues

SUMMARY:
Somatic mutations in the MAP (mitogen-activated protein) kinase pathway have been found in about 80% of papillary thyroid tumors (PTCs). The evaluation of the PTC mutational profile is crucial for the definition of the prognosis and for predicting the effects of targeted and personalized therapies. Molecular characterization by mass spectrometry (Mass ARRAY) allows the search for multiple mutations in a single experiment, in a sensitive, fast and economic way. A Mass ARRAY platform (PTC-MA) was developed, capable of identifying the presence of the most common somatic point mutations and rearrangements in PTC (Pesenti et al., Endocrine 2017). The aim of the study is to characterize the mutational profile of a large series of papillary thyroid carcinomas (PTC). Tumor samples will be analyzed using our PTC-MA platform. The molecular profile of PTCs will be correlated with the clinical and prognostic characteristics of the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with papillary thyroid cancer
* patients whose tumor tissue can be recovered for genetic analysis

Exclusion Criteria:

* patients who did not give consent
* patients lost to follow-up
* tumor samples not suitable for genetic analysis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with papillary thyroid cancer, operated and followed by our Center of Excellence for the Diagnosis and Treatment of Thyroid Tumors
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mutational profile of PTCs | years 1-8
  The mutational profile of about 600 PTCs will be characterized and correlate with the clinical characteristics and patient outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Laura Fugazzola, MD PhD, Principal Investigator — Istituto Auxologico Italiano-Milan, Italy
Locations (1):
- Istituto Auxologico Italiano, Milan, MI, Italy

REFERENCES:
- [Result] Pesenti C, Muzza M, Colombo C, Proverbio MC, Fare C, Ferrero S, Miozzo M, Fugazzola L, Tabano S. MassARRAY-based simultaneous detection of hotspot somatic mutations and recurrent fusion genes in papillary thyroid carcinoma: the PTC-MA assay. Endocrine. 2018 Jul;61(1):36-41. doi: 10.1007/s12020-017-1483-2. Epub 2017 Dec 6. PMID 29214440